CLINICAL TRIAL: NCT03134677
Title: The Effects of Different Anesthetic Techniques on QT, Corrected QT (QTc), and P Wave Dispersions in Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sevtap Hekimoglu Sahin, Clinical Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUTF-GOKAEK 2014/116
Record Dates: First submitted 2017-03-30; First posted 2017-05-01 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Caesarean Section; Anesthesia; Reaction
Keywords: Spinal anesthesia; General anesthesia; P wave dispersion
MeSH Terms: interventions — Bupivacaine; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Bupivacaine (Experimental): We were performed spinal anesthesia sitting position by midline. After confirming the free flow of cerebrospinal fluid, bupivacaine was administered without aspiration.ECG recordings were performed at preoperative, 5, 15, and 30 minutes after initial anesthesia and 30 minutes post-operatively.
  Interventions: Drug: Bupivacaine
- Sevoflurane (Experimental): We were performed general anesthesia with sevoflurane. Anesthesia was maintained with 2-3% sevoflurane. ECG recordings were performed at preoperative, 5, 15, and 30 minutes after initial anesthesia and 30 minutes post-operatively.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Bupivacaine — 2 ml of hyperbaric bupivacaine (0.5%) was given intrathecally to patients in a sitting position by midline attempt between the L3 and L4 intervertebral space.ECG recordings were performed at preoperative, 5, 15, and 30 minutes after initial anesthesia and 30 minutes post-operatively.
  Other Names: Marcaine Heavy 0.5%
  Arms: Bupivacaine
Drug: Sevoflurane — General anesthesia was maintained with 2-3% sevoflurane. ECG recordings were performed at preoperative, 5, 15, and 30 minutes after initial anesthesia and 30 minutes post-operatively.
  Other Names: Sevofluran
  Arms: Sevoflurane

SUMMARY:
This study evaluates the effects of different anesthetic techniques on QT, QTc, and Pwd in cesarean section. Half of participants received general anesthesia, while the other half received spinal anesthesia Electrocardiography (ECG) recordings were performed at preoperative, 5, 15, 30 min after initiation anesthesia and 30 min post-operatively. Hemodynamic state were also recorded at the same time intervals. QT, corrected QT (QTc), QT dispersion (QTd), QTc dispersion (QTcd), P-wave dispersion (Pwd), corrected JT interval, T wave (Tp-e), transmular dispersion of repolarization durations were measured from ECG records at predetermined time intervals of spinal or general anesthesia.

DETAILED DESCRIPTION:
The anesthetic drugs used according general or regional anesthesia techniques can display proarrhythmic and antiarrhythmic effects by inducing cardiac electrical signals with different pathways.In addition, comorbid disease, hormonal changes, surgery procedures, and drug therapy can all cause arrhythmia in the intraoperative period. Likewise, pregnancy causes many changes hormonal and physiological in women. Hemodynamic and hormonal changes during pregnancy can cause effects proarrhythmogenic that cause premature atrial and ventricular beats to develop.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists physical status I-II
2. ages 20-40 years
3. parturient patients

Exclusion Criteria:

1. spinal cord and peripheral nervous system diseases;
2. hypovolemic and hemorrhagic shock;
3. increased intracranial pressure;
4. severe anemia;
5. systemic infection;
6. scoliosis;
7. congenital spinal anomalies;
8. vertebral colon metastatic lesions;
9. anticoagulant drug use;
10. diabetes mellitus;
11. hypo/hyperthyroidism;
12. atrial and/or ventricular hypertrophy on ECG;
13. cardiomyopathy;
14. valvular disease;
15. cardiac failure or chronic disease;
16. cardiomegaly
17. used medication causing QT interval prolongation.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — elective cesarean section
Enrollment: 90 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2016-07-23 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
Measurement of perioperative electrocardiogram changes | Preoperative, intraoperative and postoperative 30 min.
  Electrocardiography measurements were performed and recorded for patients at preoperative, intraoperative 5th, 15th, 30th minutes and postoperative 30th minutes. Electrocardiogram is assessed change from Baseline at intraoperative and postoperative 30 min. Treatment-Related Adverse Events, cardiac disorder Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Sevtap Hekimoglu Sahin, Professor, Study Director — Trakya University Medical Faculty

IPD SHARING:
Plan to Share IPD: Undecided